CLINICAL TRIAL: NCT05217381
Title: Retrospective Observational Study With Real-World Data to Assess Demographic and Clinicopathological Profiles, and Management of Breast Cancer Patients With Positive, Low or Negative Expression of HER2 in Spain
Brief Title: Real-World Data of Clinicopathological Characteristics and Management of Breast Cancer Patients According to HER2 Status
Acronym: RosHER
Status: Completed | Type: Observational
Sponsor: MedSIR (Other)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MEDOPP367
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Early Breast Cancer; Metastatic Breast Cancer; Locally Advanced Breast Cancer
Keywords: Breast Cancer; Real-World Data; HER2 negative; HER2 positive; HER2 low; Artificial Intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with an initial diagnostic of early breast cancer or locally advanced breast cancer or de novo metastatic breast cancer

SUMMARY:
This is a data-driven, retrospective, longitudinal, population- based, observational, multi-centered study using secondary data captured from congruent electronic health records (EHRs).

DETAILED DESCRIPTION:
Patients with pathologically documented an initial breast cancer diagnostic (early breast cancer (BC) or locally advanced BC or de novo metastatic BC) with documented human epidermal growth factor receptor 2 (HER2) and estrogen receptor (ER)/progesterone receptor (PgR) expression status at the time of diagnosis.

Data to determine the primary endpoint is estimated to be derived from the EHRs of over 2,000 patients that have an initial diagnosis of early BC, or locally advanced BC, or de novo metastatic BC (mBC) between the 1st of January 2005 and the 31st of December 2021, and who had at least one subsequent relapse until the 31st of December 2021 in at least 10 clinical centers.

The secondary endpoints utilize a larger collection of data from over 30,000 patients that have an initial diagnosis of early BC, or locally advanced BC, or de novo mBC between the 1st of January 2005 and the 31st of December 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who have at least 18 years of age at enrollment.
2. Patients with initial diagnosis of early BC or locally advanced BC or de novo mBC between the 1st of January 2005 and the 31st of December 2021
3. Pathologically documented BC for:

   * HER2 receptor expression with a validated assay according to American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) recommendations at the time of diagnosis. HER2 receptor expression can be: o HER2-positive expression: defined as immunohistochemistry (IHC) 3+ or concurrent IHC 2+ with in situ hybridization (ISH) positive or HER2-low expression: defined as IHC 2+ with ISH-negative or IHC 1+ with ISH-negative or untested) or HER2-negative expression: defined as IHC: 0.
   * Estrogen receptor [ER]- and/or progesterone receptor [PgR] with a validated assay according to ASCO/CAP guidelines at the time of diagnosis during early and/or advanced setting. ER/PgR expression can be: positive: ER or PgR ≥1% or negative: ER and PgR <1%
4. Electronic Health Records (EHRs), with guaranteed data to meet requisites, about clinicopathological characteristics, type of surgery, treatment management, disease outcomes, and genomic profile. Centers that agree to participate must commit to include all subjects who meet the inclusion criteria, in order to reduce possible selection bias.

Exclusion criteria:

1. Medical charts at Hospital that cannot guarantee reliable and congruent EHRs.
2. If sufficient data cannot be obtained from EHRs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an initial confirmed diagnostic of breast cancer (early or locally advanced or de novo metastatic) managed in clinical practice during the predefined timeframe in the selected hospitals.
Sampling Method: Probability Sample
Enrollment: 18533 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of HER2 expression change between initial diagnosis versus any of the subsequent BC relapses | 180 months
  Change in HER2 expression between initial diagnosis of early BC or locally advanced BC or de novo mBC and any of subsequent BC relapses by IHC and/or ISH validated assays.

SECONDARY OUTCOMES:
Prevalence of changes in HER2 expression among different lines of treatment | 180 months
  HER2 expression changes as assessed by IHC (0+, 1+, 2+, 3+) and/or ISH (positive or negative) validated assays among different lines of treatment in the advanced setting, and/or among different metastatic sites.
Description of the clinicopathological characteristics | 180 months
  Description of all the comprehensive clinicopathological characteristics (age at diagnosis, gender [male or female], baseline Eastern Cooperative Oncology Group [ECOG] performance status [0, 1, or 2], breast cancer pathological subtype at primary site, intrinsic subtype at primary and/or metastatic site by PAM50 test [including luminal A, luminal B, HER2-overexpressing, and basal-like], ER and PgR status [positive and/or negative] at primary and/or metastatic site, HER2 status by IHC and/or ISH testing [HER2-positive, HER2-low expressing, and HER2-negative status per ASCO-CAP guidelines] at primary and/or metastatic site, Ki67 at primary and/or metastatic site, endocrine resistance [primary or secondary]), metastatic sites (bone, brain, visceral involvement) nodal involvement, presence of measurable or evaluable disease per Response Evaluation Criteria In Solid Tumors (RECIST) in all patients enrolled.
Evaluation of the disease management | 180 months
  Description of disease management and treatment patterns in all patients enrolled for gaining contemporary insights into HER2-low expressing breast cancer treatment trends that may inform clinicians for future management plans.
Description of genomic profile | 180 months
  Identification of patients' genomic profile including DNA alterations and/or RNA expression of genes commonly disrupted in breast cancer, including driver, prognostic-related, and drug-response associated genes in tissue or liquid biopsies from all patients enrolled.
Efficacy (OS) | 180 months
  Overall survival (OS) is defined as the time from date of primary treatment initiation to date of death due to any cause. In the absence of confirmation of death, survival time will be censored to last date the participant was known to be alive.
Efficacy (ORR) | 180 months
  Objective response rate (ORR) is defined as the sum of complete response (CR) and partial response (PR) relative to the number of patients in the analysis set with measurable disease at baseline as per RECIST v.1.1.
Efficacy (CBR) | 180 months
  Clinical benefit rate (CBR) is defined as the proportion of participants with CR, PR or stable disease (SD) ≥24 weeks relative to the number of patients in the analysis set as per RECIST v.1.1.
Efficacy (PFS) | 180 months
  Progression-free survival (PFS) is defined as the period of time from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using RECIST v.1.1.
Efficacy (DoR) | 180 months
  Duration of response (DoR) is defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression, death due to any cause or treatment discontinuation, whichever occurs first as per RECIST v.1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, MD, PhD, Principal Investigator — MedSIR
Locations (7):
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital Sant Joan Despí - Moisès Broggi, Barcelona
  - Hospital Universitari Son Espases, La Palma
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación de Alcorcón, Madrid
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander